CLINICAL TRIAL: NCT02586363
Title: A Randomized, Open-label, 3-way Crossover Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics and Safety of Single-dose Cavir Tab. 0.5mg With Baraclude Tab. 0.5mg in Healthy Male Volunteers
Brief Title: Study of Evaluation of Cavir Tab. 0.5mg With Food Effect on Pharmacokinetics and Safety
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Dong-seok Yim, Prof., Seoul St. Mary's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Cavir food effect study
Record Dates: First submitted 2015-10-15; First posted 2015-10-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Entecavir; Food effect; Cavir Tab 0.5mg; Baraclude Tab. 0.5mg
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baraclude Tab. 0.5mg, fasting (Active Comparator): Single dose Baraclude Tab. 0.5mg, fasting state
  Interventions: Drug: Baraclude Tab. 0.5mg, fasting
- Cavir Tab. 0.5mg, fasting (Experimental): Single dose Cavir Tab. 0.5mg, fasting state
  Interventions: Drug: Cavir Tab. 0.5mg, fasting
- Cavir Tab. 0.5mg, high fatty meal (Experimental): Single dose Cavir Tab. 0.5mg, high fatty meal
  Interventions: Drug: Cavir Tab. 0.5mg, high fatty meal

INTERVENTIONS:
Drug: Baraclude Tab. 0.5mg, fasting — After drug administration, Blood sampling for Pharmacokinetics (Entecavir concentration)
  Arms: Baraclude Tab. 0.5mg, fasting
Drug: Cavir Tab. 0.5mg, fasting — After drug administration, Blood sampling for Pharmacokinetics (Entecavir concentration)
  Arms: Cavir Tab. 0.5mg, fasting
Drug: Cavir Tab. 0.5mg, high fatty meal — After drug administration, Blood sampling for Pharmacokinetics (Entecavir concentration)
  Arms: Cavir Tab. 0.5mg, high fatty meal

SUMMARY:
In this clinical trial, the investigator will clarify the difference in pharmacokinetics between the group single dose Cavir Tab. 0.5mg and single dose Cavir Tab. 0.5mg with high fatty meal for healthy adult volunteer.

The investigators evaluate the effect of food intake on the absorption of Cavir Tab. 0.5mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, aged 19 ~ 45 at screening date
* Subject's weight is in range from -120 percentage to +120 percentage of ideal body weight which is calculated by { height (cm) - 100} * 0.9.
* The Subject is willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

* Subject has a history of clinically significant disease.
* Subject has a digestive disease (Crohn's disease, ulcer, acute or chronic pancreatitis etc) or abdomen surgery (exclude, simple appendectomy or hernia operation).
* Subject has a hypersensitivity history which is clinically significance or additives.
* Subject is inappropriate to screening (disease history, physical examination, vital sings, electrocardiogram, laboratory test etc.)
* Subject has a laboratory test result as indicated by and one of the following.

  * serum aspartate aminotransferase> 1.25 * normal limit
  * serum Total bilirubin > 1.5 * normal upper limit
  * serum CPK > 1.5 * normal upper limit
  * eGFR(estimated Glomerular Filtration Rate) calaulated by MDRD (Modification of Diet in Renal Disease) formula < 60 mL/min/1.73m2
* Subject is hypertension(SBP>140mmHg or DBP>90mmHg) or hypotension(SBP<90mmHg, DBP<60mmHg)
* Subject has a drug abusing history.
* Subject is currently abusing alcohol (more than 210 g/week), caffeine(more than 5cups/day) or smoking(more than half pack).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of Entecavir. | Within 6 Months After Final Visit of Subject
  phamacokinetic parameter
Area under the plasma concentration versus time curve, last (AUClast) of entecavir. | Within 6 Months After Final Visit of Subject.
  phamacokinetic parameter
Number of participants with adverse events. | Within 6 Months After Final Visit of Subject

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve, infinite (AUCinf) of entecavir. | Within 6 Months After Final Visit of Subject.
  Pharmacokinetic parameter
The time at which the Cmax is observed (Tmax) of entecavir. | Within 6 Months After Final Visit of Subject.
  Pharmacokinetic parameter, Cmax is the peak plasma concentration.
Terminal half-life (T1/2) of entecavir. | Within 6 Months After Final Visit of Subject.
  Pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Seok Yim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital